CLINICAL TRIAL: NCT02001597
Title: Intra-operative Trans-rectal Ultrasound Guidance for Robot-assisted Radical Prostatectomy
Acronym: TRUS-RP
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); British Columbia Innovation Council (Unknown)
Responsible Party: Principal Investigator, Septimiu E. Salcudean, Professor, University of British Columbia
Other Study IDs: H11-02267; 385902-2010 (Other Grant/Funding Number: CHRP)
Record Dates: First submitted 2013-11-22; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Prostate Cancer
Keywords: surgery; robotic; ultrasound; guidance; endorectal
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgery patients

SUMMARY:
Radical prostatectomy, or the surgical extirpation of the prostate, is a standard treatment for prostate cancer. The state of the art radical prostatectomy involves a robotic laparoscopic surgery system (the da Vinci) which provides the surgeon with excellent 3D visualization of the surgical site and improved dexterity over standard laparoscopic instruments. While the long term prognosis of prostate cancer patients who undergo radical prostatectomy has improved significantly over the past two decades, there remain significant rates of disease recurrence and complications.

The investigators hypothesis is that advanced trans-rectal ultrasound (TRUS) imaging can be deployed and used easily during surgery, can be registered to the robot coordinate systems with high accuracy, and can be controlled from the surgeon's console, in order to improve the visualization of the prostate and peri-prostatic anatomy, and in order to produce a cancer probability map that can be used to make decisions on surgical margins.

The investigators objectives are

1. To demonstrate that TRUS imaging can be integrated with the da Vinci radical prostatectomy
2. To determine the ability of TRUS imaging to intra-operatively visualize the prostate and peri-prostatic tissue from the surgical console

This is an observational study; trans-rectal ultrasound will be used to visualize the prostate and periprostatic structures during surgery but the standard of care will not be affected by this ultrasound imaging.

ELIGIBILITY:
Inclusion Criteria:

* All men who undergo robot-assisted radical prostatectomy are eligible.

Exclusion Criteria:

* None

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men who undergo robot-assisted radical prostatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Time required to register the trans-rectal ultrasound coordinates to the da Vinci coordinates | 1 year
  We will measure and report the time required to carry out the registration of the ultrasound transducer relative to the da Vinci coordinate system for each of the patients.

SECONDARY OUTCOMES:
Successful prostate visualization | 1 year
  For each patient in the cohort, we will report the total time of ultrasound use and the specific context in which it was used, e.g. identification of the bladder neck, identification of rectal wall, identification of the seminal vesicles, identification of the prostate apex.

OTHER OUTCOMES:
Impact on completion time | 1 year
  We will report the total additional ultrasound set-up time for each of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada